CLINICAL TRIAL: NCT01267513
Title: Noninvasive Ambulatory Measurements of Physiological Parameters Using a DLS-based Sensor
Brief Title: Ambulatory Measurements of Physiological Parameters
Acronym: LIFEBEAM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Collaborators: Tel Aviv University (Other)
Responsible Party: Sponsor
Other Study IDs: Oxytone/Lifebeam Monitor; MMC202/2010 (Other: Meir Hospital Center, Kfar Saba, Israel)
Record Dates: First submitted 2010-12-27; First posted 2010-12-28 (Estimated); Last update posted 2012-03-19 (Estimated); Status verified 2012-03

CONDITIONS: Non Invasive Test of Pulse and Oxygen Saturation
Keywords: oxygen saturation; pulse rate; tachycardia; bradycardia; hypoxia
MeSH Terms: conditions — Tachycardia; Bradycardia; Hypoxia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- normal volunteers: Normal individuals, aged 18 -75
- Hospitalized patients: Pulmonary and cardiac ICU, Trauma

SUMMARY:
Ambulatory monitoring of physiological variables is important in following the health status of individuals in non-hospital controlled situations. The investigators are developing a non-invasive sensor based on dynamic light scattering that is able to measure pulse, blood flow and coagulability. Oxygen saturation can also be detected with minor modification of the apparatus. The investigators plan to validate the investigators sensor by applying it to patients in the intensive care unit, or to patients undergoing cardiac stress tests. The results of the investigators sensor will not be utilized for any therapeutic decisions, but will be collected for later comparison with conventional monitoring of pulse and oxygenation with standard monitors. The monitor is worn like a wrist watch, and will collect data into a small data storage disc for later analysis.

DETAILED DESCRIPTION:
Subjects to be studied will be either individuals undergoing routine cardiac stress tests, or patients admitted to the pulmonary ward of Meir Hospital who are being monitored in conventional manner. Normal volunteers will also be tested, under the following conditions: at rest, while running, while performing calisthenics, and while crawling on the ground. If non-inferiority of the new sensor is established compared to the standard clinically used sensors, then additional studies will be performed on acutely ill patients, such as patients admitted with multi-trauma.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are able to sign informed consent.
* Patients undergoing standard cardiac stress tests who are able to sign informed consent.
* Patients with pulmonary disease who are being monitored in a routine manner who are will ing to sign informed consent.

Exclusion Criteria:

* Children
* Patients unable or unwilling to give consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Normal volunteers will be studied. Individuals undergoing routine cardiac stress testing will be studied. Stable patients admitted to the pulmanary ward who are being monitored routinely for oxygen saturation and pulse will be studied.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2011-04; Primary Completion 2012-05 (Estimated); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
Comparison of oxygen saturation and pulse rate between our sensor and conventional sensors | 0ne year
  We wish to determine non-inferiority of our new sensor compared to current non-ambulatory sensors.

CONTACTS AND LOCATIONS:
Overall Officials: Louis Shenkman, AB, MD, Principal Investigator — Meir Medicall Center
Locations (1):
- Meir Medical Center, Kfar Saba, Israel

REFERENCES:
- [Background] Shitrit D, Rusanov V, Peled N, Amital A, Fuks L, Kramer MR. The 15-step oximetry test: a reliable tool to identify candidates for lung transplantation among patients with idiopathic pulmonary fibrosis. J Heart Lung Transplant. 2009 Apr;28(4):328-33. doi: 10.1016/j.healun.2008.12.019. PMID 19332258